CLINICAL TRIAL: NCT04989140
Title: A Multi-center, Open-label, Single-arm Clinical Study of Ixazomib/Pomalidomide/Dexamethasone (IxaPD) in the Treatment of Patients With Relapsed Multiple Myeloma
Brief Title: Study of Pomalidomide, Oral Dexamethasone and Ixazomib in Patients With Relapsed MM Who Have Received Lenalidomide
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Jishuitan Hospital (Other); Beijing Chao Yang Hospital (Other); Tianjin Medical University General Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Peking University Third Hospital (Other); Beijing Hospital (Other Government); The First Affiliated Hospital of Anhui Medical University (Other); Second Hospital of Shanxi Medical University (Other); The First Affiliated Hospital of Dalian Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Junling Zhuang, Associate professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-2883
Record Dates: First submitted 2021-07-10; First posted 2021-08-04 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Multiple Myeloma
Keywords: relapsed MM; oral regiment
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- IxaPD (Experimental): Ixazomib 4 mg, capsules, orally, once on Days 1, 8 and 15 of every 28-day cycle , pomalidomide 25mg qd day 1~21 of every 28-day cycle, Dexamethasone 40 mg (20 mg for patients >75 years of age) was given on days 1, 8, 15, and 22 of every 28-day cycle.
  Interventions: Drug: Drug: Ixazomib Drug:pomalidomide Drug:dexamethasone

INTERVENTIONS:
Drug: Drug: Ixazomib Drug:pomalidomide Drug:dexamethasone — Treatment was continued until disease progression, unacceptable toxicity

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ixazomib, oral dexamethasone and in patients with relapsed multiple myeloma who have received lenalidomide.

DETAILED DESCRIPTION:
Multiple myeloma (MM), the second most common hematological malignancy, is a clonal plasma cell disorder characterized by the secretion of monoclonal immunoglobulins. The annual incidence of newly diagnosed MM (NDMM) patients is about 2-3/100,000. In the past 20 years, the median overall survival (OS) of MM patients has prolonged from 3 to 5 years to 8 to 10 years since many novel agents developed on the pipeline of treatment. For patients with relapsed/refractory multiple myeloma, the combination of new drugs can prolong the patient's progression-free survival (PFS) and overall survival (OS). At present, guidelines recommend the use of 3-4 drugs combined with chemotherapy containing proteasome inhibitors, immunomodulators or daratumomab for the treatment of patients with relapsed and refractory multiple myeloma treatment.

Bortezomib combined with lenalidomide and dexamethasone (VRd) is the first-line induction program recommended by guidelines; It has been widely used in the first-line treatment of MM patients. Therefore, when the disease relapses, the VRd regimen is not effective again. Research data shows that the second-generation oral proteasome inhibitor drug ixazomib combined with lenalidomide and dexamethasone (IxaRd) is used to treat the disease. In the treatment of RRMM patients, the progression-free survival period was significantly better than that of the lenalidomide and dexamethasone groups, and at the same time, it did not significantly increase the adverse reactions. The second-generation PI drug, Ixazomib, was approved in China in May 2018 and is widely used in RRMM patients. In addition, because most patients with multiple myeloma use lenalidomide in the first-line treatment and maintenance treatment, a large proportion of RRMM patients are resistant to lenalidomide. Pomalidomide, the third-generation oral immunomodulator drug, can overcome lenalidomide resistance and has better safety in patients with renal insufficiency MM. The results of clinical trials confirmed that pomalidomide combined with a proteasome inhibitor and dexamethasone is better than a dual-drug regimen of pomalidomide and dexamethasone in RRMM patients. A convenient and safe full oral regimen, that is, ixazomib combined with pomalidomide and dexamethasone (IxaPd) is expected to improve the efficacy and survival of RRMM patients. The purpose of this study was to evaluate the efficacy and safety of a three-drug oral regimen of ixazomib, pomalidomide and dexamethasone in patients with relapsed MM who have received lenalidomide.

At the screening visit, informed consent will be obtained from all subjects who are deemed potentially eligible for enrollment in the study, according to the protocol-specified inclusion and exclusion criteria.Eligible patients are receive treatment IxaPD. Ixazomib 4 mg, capsules, orally, once on Days 1, 8 and 15 of every 28-day cycle , pomalidomide 25mg qd day 1~21 of every 28-day cycle, Dexamethasone 40 mg (20 mg for patients >75 years of age) was given on days 1, 8, 15, and 22 of every 28-day cycle. Treatment was continued until disease progression, unacceptable toxicity.Progression free survival, overall survival, time to next treatment, overall response rate and safety issues will be recorded. Drug doses will be adjusted or withdrawn based on the degree of toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years of age or older;
2. Newly diagnosed MM patients who fulfill the diagnostic criteria of the Chinese Guidelines for the Diagnosis and Treatment of Multiple Myeloma (Revised in 2020) Standards;
3. Patients with relapsed MM who have received 1 to 3 prior therapies (including lenalidomide);
4. There must be a washout period of two weeks (14 days) from the last treatment (excluding dexamethasone treatment);
5. Previously untreated subjects with ixazomib or pomalidomide;
6. Subjects of childbearing age should take effective contraceptive measures and must agree to comply with all contraceptive requirements; Contraceptive requirements: women with fertility must decide to adopt two reliable contraceptive methods at the same time (a highly effective method of contraception-fallopian tube ligation, intrauterine contraceptive device, hormones (contraceptive pills, needles, patches, vaginal rings or implants) ) Or partner's vas deferens ligation, another effective contraceptive program-male rubber or synthetic condoms, diaphragm or cervical cap); unless the cause of hysterectomy, or a history of infertility in time, effective contraception is also required. Men must agree to use a latex condom during sexual contact with a Females of childbearing potential even if they have had a successful vasectomy;
7. Patients must have measurable disease defined by at least 1 of the following 3 measurements: Serum M-protein≥5 g/ L, Urine M-protein≥200 mg/24 hours, Serum free light chain assay: involved free light chain level≥100 mg/L, provided that the serum free light chain ratio is abnormal;
8. Hematology satisfies the following conditions: when myeloma cells are less than 50%, ANC≥1.0×109/L (including with the support of G-CSF) and PLT≥75×109/L; when myeloma cells are ≥50% , Any ANC and PLT≥50×109/L;
9. Must be able to take antithrombotic drugs, such as low molecular weight heparin sodium or aspirin;
10. Physical performance status (ECOG) score ≤ 2; Expected lifetime More than 3 months.
11. Patients participate in the study based on his/her own will and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Patients who are allergic or intolerant to ixazomib, pomalidomide or dexamethasone;
2. Patients who have used ixazomib or pomalidomide;
3. Patients who are resistant to bortezomib;
4. Patients with severe cardiopulmonary insufficiency;
5. Patients with severe liver and kidney dysfunction, ALT or AST or bilirubin exceeds 3 times the upper limit of normal range, and the creatinine clearance rate is less than 30 ml/min;
6. patients with other malignancies (except for carcinoma in situ);
7. patients with serious bacterial or viral infections, such as HIV or HBV, HCV, etc.;
8. Patients with active new thrombosis or unwilling to receive anti-thrombotic therapy;
9. Patients with extramedullary disease;
10. Patients with peripheral neuropathy ≥ Grade 3;
11. Pregnant or lactating women;
12. Can't strictly contraception;
13. Psychiatric patients and patients with other serious mental illness that potentially impact signing informed consent and disease consultation and follow-up;
14. Patients who have participated in other clinical trials within one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2024-07-26 (Estimated); Study Completion 2024-07-26 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Time Frame: From date of enrollment until the date of first documented progression, assessed up to 24 months
  From enrollment to first disease progression

SECONDARY OUTCOMES:
Adverse events assessment | Each cycle, up to 24 months of follow-up.
  Number of adverse events according to symptoms, physical examination and scheduled laboratory tests
Overall survival | At baseline, on day 1 of each cycle, and after 2, 3,4,5,7,9,11,13,16,19,22, 25 and 28 months of follow-up
  From enrollment to death with follow-up
Overall response rate | At baseline, on day 1 of each cycle, and after 2, 3,4,5,7,9,11,13,16,19,22, 25 and 28 months of follow-up
  Overall response rate included Complete Response (CR), Very good partial response (VGPR) and PR, before the new treatment, two consecutive evaluations are in line with defined criteria in order to confirm the efficacy evaluation.
Time to next treatment | At baseline, on day 1 of each cycle, and after 2, 3,4,5,7,9,11,13,16,19,22, 25 and 28 months of follow-up
  From enrollment to the time next treatment is administrated

CONTACTS AND LOCATIONS:
Overall Officials: Junling Zhuang, MD, Principal Investigator — Peking UMCH
Locations (1):
- PekingUMCH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
individual baseline characteristic ,treatment and follow-up results will be shared after publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication, the data will become available